CLINICAL TRIAL: NCT06549504
Title: An Open-label, Randomized, Fasting, Single, Oral Administration, Group 2, Stage 2, Cross-over Bioequivalence Study of AG2202 in Healthy Volunteers
Brief Title: Bioequivalence Study of AG2202
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG2202
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Bioequivalence Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AG2202T (Experimental)
  Interventions: Drug: AG2202T
- AG2202R (Active Comparator)
  Interventions: Drug: AG2202R

INTERVENTIONS:
Drug: AG2202T — AG2202T Single-dose
  Arms: AG2202T
Drug: AG2202R — AG2202R Single-dose
  Arms: AG2202R

SUMMARY:
The objective of this study is to evaluate the human bioequivalence of AG2202T and AG2202R.

DETAILED DESCRIPTION:
To evaluate the bioequivalence of two formulations of AG2202T and AG2202R after a single oral dose administration in healthy Korean subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 19 years or older at the time of screening
* Subjects with a BMI of 18.0-30.0 kg/m2
* Subjects who do not have clinically significant congenital or chronic diseases and who do not have any pathological symptoms or findings as a result of general clinical examination
* Subjects who are deemed eligible based on the screening tests

Exclusion Criteria:

* Subjects who have taken drugs that induce or inhibit drug metabolizing enzymes within 30 days prior to the first dose or who have taken drugs that may interfere with the investigational product within 10 days prior to the first dose
* Subjects who have taken the investigational drug within 6 months prior to the first dose
* Subjects who donated whole blood within 8 weeks prior to the first dose, or donated blood components within 2 weeks, or received a blood transfusion within 4 weeks prior to the first dose

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
AUC | Pharmacokinetic plasma samples collected over 36 hour period
  Area under the plasma concentration
Cmax | Pharmacokinetic plasma samples collected over 36 hour period
  Peak Plasma Concentration